CLINICAL TRIAL: NCT02207556
Title: Doxycycline to Upgrade Organ Response in Light Chain (AL) Amyloidosis (DUAL) Trial: A Phase II Open Label Study of Oral Doxycycline Administered as an Adjunct to Plasma Cell Directed Therapy in Light Chain (AL) Amyloidosis
Brief Title: Doxycycline to Upgrade Organ Response in Light Chain (AL) Amyloidosis Trial
Acronym: DUAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anita D'Souza, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22850; KL2TR001438 (NIH); K23HL141445 (NIH); 86-004-26 (Other Grant/Funding Number: American Cancer Society Institutional Research Grant)
Record Dates: First submitted 2014-07-23; First posted 2014-08-04 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Primary Systemic Amyloidosis
Keywords: AL amyloidosis; amyloidosis; light chain amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doxycycline (Experimental): Doxycycline will be administered at dose of 100mg orally twice daily for 1 year.
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Doxycycline will be continued until one of the following criteria is met:
  * Patient has completed 1 year of doxycycline therapy
  * Patient develops any grade 3-4 toxicity related to doxycycline use.
  Other Names: Doxycycline monohydrate

SUMMARY:
In this study the investigators want to find out more about the addition of the antibiotic, doxycycline, to standard anti-amyloid therapy in people with amyloidosis. The investigators want to find out whether doxycycline improves the response to standard anti-amyloid therapy and whether it causes any problems (side effects).

DETAILED DESCRIPTION:
Organ response to anti-plasma cell therapy in AL amyloidosis tends to lags behind hematologic response as chemotherapy may not clear pre-formed organ amyloid. Doxycycline has been shown to have inhibitory effects on amyloid fibril formation as well as de-fibrillogenic effects and shown to be beneficial in in vitro, murine models and other preclinical studies. The investigators will prospectively evaluate the safety and efficacy of doxycycline in AL amyloidosis patients when used in conjunction with anti-plasma cell chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy proven AL amyloidosis.
2. Patients ≥ 18 years of age are eligible.
3. Patient must provide informed consent.
4. All patients must have measurable amyloid organ involvement of a vital organ (eg. heart, liver, kidneys). Localized amyloidosis will also be eligible as long as the amyloid involvement is radiologically measurable.
5. A negative pregnancy test will be required for all women of child bearing potential. Breast feeding is not permitted.
6. Patients who have previously been taking doxycycline will be eligible as long as there is no contraindication to stay on doxycycline 100 mg twice daily (BID) for 1 year in the opinion of the treating physician.
7. Creatinine clearance of >25 ml/min.

Exclusion Criteria:

1. Patients with severe malabsorption syndrome precluding absorption of oral agents will be excluded.
2. Known intolerance or allergic reactions with doxycycline.
3. Previous chemotherapy for AL amyloidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2020-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita D'Souza, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Souza A, Szabo A, Flynn KE, Dhakal B, Chhabra S, Pasquini MC, Weihrauch D, Hari PN. Adjuvant doxycycline to enhance anti-amyloid effects: Results from the dual phase 2 trial. EClinicalMedicine. 2020 Jun 5;23:100361. doi: 10.1016/j.eclinm.2020.100361. eCollection 2020 Jun. PMID 32529175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were stratified by the type of amyloidosis. Subjects with primarily organ-based disease were classified as Localized Disease), whereas subjects with hematologic disease were classified as Systematic Disease. Each population received the same intervention but assessment of the clinical outcomes used different classification categories.
Groups:
- Doxycycline (Localized Disease); Doxacycline (Systemic Disease): Doxycycline will be administered at dose of 100mg orally twice daily for 1 year.
  Doxycycline: Doxycycline will be continued until one of the following criteria is met:
  * Patient has completed 1 year of doxycycline therapy
  * Patient develops any grade 3-4 toxicity related to doxycycline use.
Period: Overall Study
Arm/Group | Doxycycline (Localized Disease) | Doxacycline (Systemic Disease)
Started | 7 | 25
Completed | 5 | 20
Not Completed | 2 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 5

BASELINE CHARACTERISTICS:
Population: Two subjects in the Localized Disease arm signed consent, but did not proceed to the treatment phase of the study. One subject withdrew consent and one subject was determined to be ineligible and was withdrawn by the investigator. Baseline demographic data were collected for these subjects.
Groups:
- Doxycycline (Systemic Disease): Doxycycline will be administered at dose of 100mg orally twice daily for 1 year.
  Doxycycline: Doxycycline will be continued until one of the following criteria is met:
  * Patient has completed 1 year of doxycycline therapy
  * Patient develops any grade 3-4 toxicity related to doxycycline use.
- Total: Total of all reporting groups
Arm/Group | Doxycycline (Localized Disease) | Doxycycline (Systemic Disease) | Total
Number analyzed (Participants) | 7 | 25 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 16 | 19
  >=65 years | 4 | 9 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.6) | 65.5 (11.4) | 62.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 2 | 16 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 25 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 7 | 21 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 25 | 32

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Response
Description: This measure will record the number of subjects for each grade of response to therapy for subjects with Systematic Disease (hematologic) only. Hematologic response will be determined as follows.
  Complete response (CR) - Negative serum/urine immunofixation with normal Free Light Chain (FLC) ratio
  Very Good Partial Response (VGPR)- Difference between involved and uninvolved FLCs (dFLC) < 40 mg/L
  Partial Response (PR)- dFLC decrease > 50%
  No Response (NR)- less then PR.
Time Frame: 1 year
Population: Hematologic response is not relevant to subjects with localized disease. Subjects with localized disease were not included in this analysis. Five participants had expired by the 1 year time point
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline (Systemic Disease)
Number analyzed (Participants) | 25
Participants
  Complete Response (CR) | 6
  Partial Response (PR) | 3
  Very Good Partial Response (VGPR) | 11
  Expired at 1 year | 5

2. Secondary Outcome: Amyloid Organ Response
Description: This measure is the number of subjects (systemic disease only) for each grade of response. Efficacy will be measured in heart, liver, or kidney.
  Heart N-terminal (NT)-proBNP response >30% and > 300 ng/L decrease in patients with baseline NT-proBNP ≥650 ng/L (Patients with progressively worsening renal function cannot be scored for NT-proBNP progression).
  Improvement by 2 New York Heart Association (NYHA) classes without an increase in diuretic use or in echocardiographic wall thickness ≥ 2 mm reduction in the interventricular septal thickness by echocardiogram or improvement of ejection fraction by ≥20%.
  Liver
  ≥50% decrease in an initially elevated alkaline phosphatase level, or Decrease in liver size by at least 2 cm by ultrasound.
  Kidney 50% reduction in 24-hour urine protein excretion (at least 0.5 g/day) without worsening of creatinine or creatinine clearance by 25% over baseline.
  Soft Tissue RECIST criteria will be used.
Time Frame: 6 months and 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Doxycycline (6 Months); Doxycycline (1 Year): Doxycycline will be administered at dose of 100mg orally twice daily for 1 year.
  Doxycycline: Doxycycline will be continued until one of the following criteria is met:
  * Patient has completed 1 year of doxycycline therapy
  * Patient develops any grade 3-4 toxicity related to doxycycline use.
Arm/Group | Doxycycline (6 Months) | Doxycycline (1 Year)
Number analyzed (Participants) | 25 | 25
Participants
  Progressive Disease | 8 | 3
  Stable Disease | 8 | 8
  Response | 6 | 9
  Expired | 3 | 5

3. Secondary Outcome: Mortality
Description: The number of living subjects will be determined at Baseline, 3 months, 6 months and 1 year
Time Frame: Baseline, 3 months, 6 months, 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline (Localized Disease) | Doxacycline (Systemic Disease)
Number analyzed (Participants) | 6 | 25
Participants
  Baseline | 6 | 25
  3 Months | 6 | 23
  6 Months | 6 | 22
  1 Year | 6 | 20

4. Secondary Outcome: Patient-reported Health Quality of Life
Description: Subjects will complete the Patient Reported Outcomes Measurement Information System Global Health instrument, a 10-item standardized patient-reported outcome measure that provides global ratings of physical function, fatigue, pain, emotional distress to report on common domains of health-related quality of life. The survey comprises a series of 5-response Likert-style questions. For each question, a low score indicates lesser or absent symptom or condition and higher indicates more severe symptom or condition (e.g., 1= None to 5=Very severe). Automated scoring produces a T-score for each domain. This measure reports the physical health score. T-scores for this domain range from 16.2 to 67.7. Higher scores indicate poorer physical health.
Time Frame: Baseline, 3, 6, 9 and 12 months
Population: One subject in the Localized cohort withdrew consent prior to the 6-month visit. Five subjects in the Systemic Disease cohort expired during the course of the study; two subjects came off study; and one was lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Doxycycline (Localized Disease) | Doxacycline (Systemic Disease)
Number analyzed (Participants) | 6 | 25
score on a scale
  Baseline | 46.1 (9.4) | 40.9 (0.3)
  3 Months: number analyzed (Participants) | 6 | 22
  3 Months | 51.1 (8.8) | 40.2 (0.4)
  6 Months: number analyzed (Participants) | 5 | 20
  6 Months | 48.3 (6.3) | 40.6 (0.4)
  9 Months: number analyzed (Participants) | 5 | 20
  9 Months | 48.9 (8.0) | 41.7 (0.5)
  12 Months: number analyzed (Participants) | 5 | 17
  12 Months | 49.4 (7.7) | 44.3 (0.4)

5. Secondary Outcome: Patient-reported Mental Quality of Life
Description: Subjects will complete the Patient Reported Outcomes Measurement Information System Global Health instrument, a 10-item standardized patient-reported outcome measure that provides global ratings of physical function, fatigue, pain, emotional distress to report on common domains of health-related quality of life. The survey comprises a series of 5-response Likert-style questions. For each question, a low score indicates lesser or absent symptom or condition and higher indicates more severe symptom or condition (e.g., 1= None to 5=Very severe). Automated scoring produces a T-score for each domain. This measure reports the mental health score. T-scores for this domain range from 21.2 to 67.6. Higher scores indicate poorer mental health.
Time Frame: Baseline, 3, 6, 9 and 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Doxycycline (Localized Disease) | Doxacycline (Systemic Disease)
Number analyzed (Participants) | 6 | 25
score on a scale
  Baseline | 52.1 (10.4) | 47.9 (0.6)
  3 Month: number analyzed (Participants) | 6 | 22
  3 Month | 51.4 (10.0) | 46.0 (0.5)
  6 Months: number analyzed (Participants) | 5 | 20
  6 Months | 51.2 (9.0) | 46.4 (0.5)
  9 Months: number analyzed (Participants) | 5 | 20
  9 Months | 52.6 (11.9) | 46.7 (0.5)
  12 Months: number analyzed (Participants) | 5 | 17
  12 Months | 50.7 (10.2) | 50.6 (0.6)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Grade was determined using the Common Terminology Criteria for Adverse Events (CTCAE) v 4.03. Events graded as 4 or 5 were considered serious regardless of the standard criteria.
Arm/Group | Doxycycline (Localized Disease) | Doxycycline (Systemic Disease)
All-Cause Mortality (participants affected / at risk) | 0/5 | 5/25
Serious Adverse Events (participants affected / at risk) | 1/5 | 13/25
Other Adverse Events (participants affected / at risk) | 5/5 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline (Localized Disease) (N=5) | Doxycycline (Systemic Disease) (N=25)
Lymphocyte production decreased (Blood and lymphatic system disorders) | 0 (0) | 7 (7) — CTCAE v4.03 Grade 4
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 0 (0) | 6 (6) — CTCAE v4.03 Grade 4
Platelet Count Decreased (Blood and lymphatic system disorders) | 0 (0) | 10 (10) — CTCAE v4.03 Grade 4
White Blood Cell Count Decreased (Blood and lymphatic system disorders) | 0 (0) | 5 (5) — CTCAE v4.03 Grade 4
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 4
Adenovirus Infection (Infections and infestations) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 4
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 4
Progressive cardiac amyloidosis (Cardiac disorders) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 5
Death in Hospice (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 5
Natural Death (Cardiac disorders) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 5
Thrombosis of Vein of Lower Limb (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 4
Aspartate Aminotransferase Increased (Hepatobiliary disorders) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 4
Alanine Aminotransferase Increased (Hepatobiliary disorders) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 4
Bacterial Sepsis (Infections and infestations) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 4
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — CTCAE v4.03 Grade 4
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — CTCA v4.03 Grade 5
Drug-Induced Lupus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — CTCAE v4.03 Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline (Localized Disease) (N=5) | Doxycycline (Systemic Disease) (N=25)
Fatigue (General disorders) | 3 (3) | 15 (15)
Hypertension (Vascular disorders) | 3 (3) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 12 (12)
Edema, Limb (General disorders) | 2 (2) | 15 (15)
Hypercalcemia (Investigations) | 2 (2) | 6 (6)
Hyperglycemia (Investigations) | 2 (2) | 17 (17)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Investigations) | 2 (2) | 16 (16)
Nausea (Gastrointestinal disorders) | 2 (2) | 14 (14)
Pain (General disorders) | 2 (2) | 8 (8)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 11 (11)
Anxiety (Psychiatric disorders) | 1 (1) | 8 (8)
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cardiac Tropinin T Increased (Cardiac disorders) | 1 (1) | 4 (4)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 12 (12)
Depression (Psychiatric disorders) | 1 (1) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 15 (15)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 9 (9)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperkalemia (Investigations) | 1 (1) | 7 (7)
Hypoalbuminemia (Investigations) | 1 (1) | 15 (15)
Hypokalemia (Investigations) | 1 (1) | 14 (14)
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Low Vitamin D (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lung Crackles (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 11 (11)
Paresthesia (Nervous system disorders) | 1 (1) | 6 (6)
Rhinitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Rib Pain (General disorders) | 1 (1) | 0 (0)
Streptococcal Test, Positive (Infections and infestations) | 1 (1) | 0 (0)
Sunburn (Burn) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urine Output Decreased (Renal and urinary disorders) | 1 (1) | 0 (0)
Weight Gain (Investigations) | 1 (1) | 6 (6)
Weight Loss (Investigations) | 1 (1) | 16 (16)
Platelet Count Decreased (Investigations) | 0 (0) | 8 (8)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 12 (12)
White Cell Count Decreased (Investigations) | 1 (1) | 10 (10)
Neutrophil Cound Decreased (Investigations) | 0 (0) | 6 (6)
AST Increased (Investigations) | 1 (1) | 8 (8)
ALT Increased (Investigations) | 1 (1) | 5 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 15 (15)
Dizziness (Nervous system disorders) | 0 (0) | 15 (15)
Dysgeusia (Nervous system disorders) | 0 (0) | 13 (13)
Insomnia (Psychiatric disorders) | 0 (0) | 13 (13)
Constipation (Gastrointestinal disorders) | 0 (0) | 11 (11)
Hypotension (Vascular disorders) | 0 (0) | 11 (11)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 10 (10)
Creatinine Increased (Investigations) | 0 (0) | 10 (10)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (10)
Hypocalcemia (Investigations) | 0 (0) | 10 (10)
Tachycardia (Cardiac disorders) | 0 (0) | 9 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8)
Fever (General disorders) | 0 (0) | 8 (8)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 8 (8)
Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 7 (7)
Bloating (Gastrointestinal disorders) | 0 (0) | 7 (7)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 7 (7)
Headache (Nervous system disorders) | 0 (0) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Noncardiac Chest Pain (General disorders) | 0 (0) | 7 (7)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Hyopohosphatemia (Investigations) | 0 (0) | 6 (6)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 6 (6)
Sore Throat (Gastrointestinal disorders) | 0 (0) | 6 (6)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 6 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (6)
Chills (General disorders) | 0 (0) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Hypomagnesemia (Investigations) | 0 (0) | 5 (5)
Proteinuria (Renal and urinary disorders) | 0 (0) | 5 (5)
Bilirubin Increased (Investigations) | 0 (0) | 4 (4)
Hematuria (Renal and urinary disorders) | 0 (0) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 4 (4)
Left Atrium Enlarged (Cardiac disorders) | 0 (0) | 4 (4)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Palpitations (Cardiac disorders) | 0 (0) | 4 (4)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Blurred Vison (Eye disorders) | 0 (0) | 3 (3)
Chest Pain - Cardiac (Cardiac disorders) | 0 (0) | 3 (3)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3)
Gait Disturbance, Unsteady (General disorders) | 0 (0) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypermagnesemia (Investigations) | 0 (0) | 3 (3)
Irregular Heartbeat (Cardiac disorders) | 0 (0) | 3 (3)
Jugular Vein Distention (Vascular disorders) | 0 (0) | 3 (3)
Macroglossia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Mucocitis, Oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Periorbital Edema/Puffiness (Eye disorders) | 0 (0) | 3 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Right Atrium Enlarged (Cardiac disorders) | 0 (0) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 3 (3)
Akathisia (Nervous system disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Chest Tightness (Cardiac disorders) | 0 (0) | 2 (2)
Cyanosis (Vascular disorders) | 0 (0) | 2 (2)
Dry Eye (Eye disorders) | 0 (0) | 2 (2)
Edema, Tongue (General disorders) | 0 (0) | 2 (2)
Erythematous Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eye Discharge (Eye disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flushiing (Vascular disorders) | 0 (0) | 2 (2)
Hypernatremia (Investigations) | 0 (0) | 2 (2)
Hypersomnia (Nervous system disorders) | 0 (0) | 2 (2)
Hypoglycemia (Investigations) | 0 (0) | 2 (2)
Inguinal Hernia Repair (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Injury to Lip (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Murmur, Systolic II/IV (Cardiac disorders) | 0 (0) | 2 (2)
Night Sweats (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Petichial Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 0 (0) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Skin Tear (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Thrush (Infections and infestations) | 0 (0) | 2 (2)
Ulceration, Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary Urgency (Renal and urinary disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Watering Eyes (Eye disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT02207556/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT02207556/ICF_001.pdf